CLINICAL TRIAL: NCT04742361
Title: Phase III Study of [18F]PSMA-1007 Positron Emission Tomography for the Detection of Prostate Cancer Lesions in Patients With Biochemical Recurrence After Previous Definitive Treatment for Localized Prostate Cancer
Brief Title: Efficacy of [18F]PSMA-1007 PET/CT in Patients With Biochemial Recurrent Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ABX advanced biochemical compounds GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ABX-CT-303
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Prostate Cancer Recurrent
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F]PSMA-1007 (Experimental): single intravenous administration of [18F]PSMA-1007 for Positron Emission Tomography (PET) scan
  Interventions: Drug: [18F]PSMA-1007

INTERVENTIONS:
Drug: [18F]PSMA-1007 — diagnostic radiopharmaceutical for PET scan

SUMMARY:
This study evaluates the diagnostic performance and safety of [18F]PSMA-1007 PET/CT imaging in patients with suspected recurrence of prostate cancer after previous definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male with original diagnosis of adenocarcinoma of the prostate with prior definitive therapy
* Suspicion of recurrence or persistence

  * after radiotherapy or cryotherapy: 3 consecutive PSA rises and/or PSA rise by 2.0 ng/mL or more above nadir (ASTRO-Phoenix)
  * after prostatectomy, PSA > 0.2 ng/mL on 2 or more determinations (recurrence), or failure of PSA to fall to undetectable levels post-prostatectomy (persistence) (American Urological Association)
* For patients who previously had radical prostatectomy, salvage radiotherapy is one likely treatment plan; for patients who initially underwent radiotherapy (including brachytherapy), confirmation of low volume disease is needed to define (local) treatment.
* Life expectancy of 6 months or more as judged by the investigator
* Willing and able to undergo all study procedures
* Informed consent in writing

Exclusion Criteria:

* Age: less than18 years
* Contraindications to any of the ingredients of [18F]PSMA-1007
* Close affiliation with the investigational site
* At the time of enrolment into this study, participating in another therapeutic clinical trial or has completed study participation in another therapeutic clinical trial within 5 days of enrolment into this trial
* Having been previously enrolled in this clinical trial
* Mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial
* Being clinically unstable or requiring emergency treatment
* Patients who are unwilling to consider a biopsy if clinically recommended
* Patients who are unable to undergo a PET/CT scan
* Patients for whom systemic therapy is the most likely course regardless of PET findings.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Region-level positive predictive value (PPV) of [18F]PSMA-1007 using a combined standard of truth (SOT) | Within 6 months after PET/CT
Patient-level correct detection rate of [18F]PSMA-1007 | Within 6 months after PET/CT

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer Center, Houston, Texas
  - Excel Diagnostics and Nuclear Oncology Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- RUMC, Nijmegen, Netherlands
- Inselspital, Universitätsspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No